CLINICAL TRIAL: NCT05263219
Title: Transarterial Chemoembolization With Drug-eluting Beads Plus Hepatic Arterial Infusion Chemotherapy Versus Hepatic Arterial Infusion Chemotherapy Alone for Large Hepatocellular Carcinoma
Brief Title: DEB-TACE+HAIC vs. HAIC for Large HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Hainan General Hospital (Other); Maoming People's Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); Affiliated Hospital of Guangdong Medical University (Other); First People's Hospital of Foshan (Other); Jiangmen Central Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-09
Record Dates: First submitted 2022-02-12; First posted 2022-03-02 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Transarterial chemoembolization; Hepatic arterial infusion chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transarterial chemoembolization with drug-eluting beads plus hepatic arterial infusion chemotherapy (Experimental): Patients will receive the combination treatment of DEB-TACE and HAIC.
  Interventions: Procedure: dTACE-HAIC; Drug: dTACE-HAIC protocol
- Hepatic arterial infusion chemotherapy (Active Comparator): Patients will receive HAIC treatment alone.
  Interventions: Procedure: HAIC; Drug: HAIC protocol

INTERVENTIONS:
Procedure: dTACE-HAIC — For DEB-TACE, superselective catheterization is performed and CalliSpheres loaded with pirarubicin is use for chemoembolization. The embolization end point was blood stasis of the tumor-feeding arteries. In patients with huge or bilobar multiple lesions, in order to reduce the risk of complications, the embolization end point was not achieved in the initial TACE but in the second or third TACE session.
  After each chemoembolization, the microcatheter is reserved at the proper/left/right hepatic artery. The FOLFOX-based regimen is intra-arterially administered.
  During follow-up, the treatment will be repeated on demand (at a 4-6-week interval usually) based on the evaluation of the follow-up laboratory and imaging examination.
  Arms: Transarterial chemoembolization with drug-eluting beads plus hepatic arterial infusion chemotherapy
Procedure: HAIC — HAIC treatment is divided into 3-week cycles. The microcatheter is advanced into the proper/left/right hepatic artery on day 1 in every cycle of treatment. After the patient returned to the ward, the FOLFOX-based regimen is intra-arterially administered though the microcatheter.
  The treatment is repeated once every 3 weeks for up to six cycles.
  Arms: Hepatic arterial infusion chemotherapy
Drug: dTACE-HAIC protocol — CalliSpheres (100-300 µm) loaded with pirarubicin for transarterial chemombolization: Typically, one vial of the beads was loaded with 60 mg pirarubicin. If blushed tumors is still visible after the embolization with one vial of beads, regular microspheres (8spheres) with diameters of 100-700 μm are additionally injected.
  FOLFOX-based regimen for hepatic arterial infusion chemotherapy: oxaliplatin, 85 mg/m2 infusion for 2 hours; leucovorin, 400 mg/m2 infusion for 2 hours; and 5-FU, 400 mg/m2 bolus infusion and then 2400 mg/m2 continuous infusion over 46 h.
  Other Names: Drugs for DEB-TACE and HAIC
  Arms: Transarterial chemoembolization with drug-eluting beads plus hepatic arterial infusion chemotherapy
Drug: HAIC protocol — FOLFOX-based regimen for hepatic arterial infusion chemotherapy: oxaliplatin, 85 mg/m2 infusion for 2 hours; leucovorin, 400 mg/m2 infusion for 2 hours; and 5-FU, 400 mg/m2 bolus infusion and then 2400 mg/m2 continuous infusion over 46 h.
  Other Names: Drugs for HAIC
  Arms: Hepatic arterial infusion chemotherapy

SUMMARY:
This study is conducted to evaluate the efficacy and safety of transarterial chemoembolization with drug-eluting beads (DEB-TACE) plus hepatic artery infusion chemotherapy (HAIC) compared with HAIC alone for unresectable large hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a multicenter, prospective and randomized study to evaluate the efficacy and safety of DEB-TACE (with CalliSpheres) plus HAIC compared with HAIC alone for unresectable large HCC (>7cm).

230 patients with initially unresectable large HCC (> 7cm) will be enrolled in this study. The patients will receive either DEB-TACE plus HAIC (dTACE-HAIC) or HAIC as the primary treatment using an 1:1 randomization scheme. In the dTACE-HAIC arm, the microcatheter will be reserved at the proper/left/right hepatic artery and chemotherapy drugs (FOLFOX-based regimen) will be intra-arterially administered though the microcatheter. The treatment can be repeated on demand (at a 4-6-week interval usually) based on the evaluation of follow-up laboratory and imaging examination by the multidisciplinary team. In the HAIC arm, treatment will repeated once every 3 weeks for up to six cycles. During follow-up, the potential resectability of the tumor will be assessed by the multidisciplinary team (MDT). Once the tumors become resectable, curative surgical resection will be recommended for the patients.

The primary end point of this study is overall survival (OS). The secondary endpoints are tumor response (objective response rate and disease control rate), success rate of conversion to resection, progression-free survival (PFS), and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC confirmed by histology/cytology or diagnosed clinically.
* The maximum HCC lesion > 7 cm.
* Unresectable HCC evaluated by the surgeon team.
* At least one measurable intrahepatic target lesion.
* Patients without cirrhosis, or with cirrhosis but the liver function of Child-Pugh Class A.
* ECOG score of performance status ≤ 1 point.
* Adequate organ and bone marrow function; the blood biochemical examination: platelet count ≥75×10^9/L, leukocyte >3.0×10^9/L, ASL and AST≤5×ULN, creatinine≤1.5×ULN, INR<1.5 or PT/APTT normal range.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Accompanied with tumor thrombus involving the main portal vein or bilateral first-order branch of portal vein.
* Accompanied with vena cava tumor thrombus.
* Extrahepatic metastasis.
* Previous treatment with TACE, HAIC, liver transplantation, resection, ablation, radiotherapy, or systemic therapy.
* Decompensated liver function, including: ascites, bleeding from gastroesophageal varices, and hepatic encephalopathy.
* Those with organs (heart and kidneys) dysfunction who cannot tolerate TACE or HAIC treatment.
* History of other malignancies.
* Uncontrollable infection.
* History of HIV.
* Allergic to the drugs involved in the research.
* Patients with gastrointestinal bleeding within 30 days, or other bleeding> CTCAE grade 3.
* History of organ or cells transplantation.
* Those with bleeding tendency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 4 years.
  The time from date of randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) per mRECIST. | 4 years.
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to mRECIST.
ORR per RECIST 1.1. | 4 years.
  The proportion of patients with the best response of CR or PR according to RECIST 1.1.
Disease control rate (DCR) per mRECIST. | 4 years.
  The proportion of patients with the best response of CR, PR, or stable disease (SD) according to mRECIST.
DCR per RECIST 1.1. | 4 years.
  The proportion of patients with the best response of CR, PR, or SD according to RECIST 1.1.
Progression free survival (PFS) per mRECIST. | 4 years.
  The time from date of randomization until the first occurrence of disease progression (according to mRECIST) or death due to any cause, whichever occurs first.
Progression free survival (PFS) per RECIST 1.1. | 4 years.
  The time from date of randomization until the first occurrence of disease progression (according to RECIST 1.1) or death due to any cause, whichever occurs first.
Success rate of conversion to resection | 4 years.
  The proportion of patients with initially unresectable large HCC who were evaluated by the surgical team as suitable for surgical resection after dTACE-HAIC or HAIC treatment.
Adverse Events (AEs) | 4 years.
  Number of patients with AEs assessed by Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Kangshun Zhu, Dr., Study Chair — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China